CLINICAL TRIAL: NCT00721227
Title: Assessment of Gastric Volume Reduction in Surgical Weight Loss Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Amy Mahanes, Senior Clinical Research Associate, Ethicon Endo-Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-07-0005
Record Dates: First submitted 2008-07-09; First posted 2008-07-24 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior Curve (Active Comparator): Reduction Gastroplasty by Gastric Plication on Anterior Curve
  Interventions: Procedure: Reduction Gastroplasty
- Greater Curve (Active Comparator): Reduction Gastroplasty by Gastric Plication on Greater Curve
  Interventions: Procedure: Reduction Gastroplasty

INTERVENTIONS:
Procedure: Reduction Gastroplasty — * Subjects will undergo reduction gastroplasty by gastric plication
  * Subjects are followed for 12 months to evaluate outcomes and potential complications.

SUMMARY:
This trial will assess the feasibility of reduction gastroplasty with standard suture in bariatric patients who are candidates for surgical weight loss intervention.

DETAILED DESCRIPTION:
The overall plan for all subjects consists of the following elements:

* Subject will be informed about the nature of the research, given the Informed Consent Document (ICD) to read, and if the subject understands and agrees to the procedure will be asked to sign a written informed consent (the ICD).
* Subjects will undergo reduction gastroplasty by gastric plication in which a section of the stomach will be infolded by multiple rows of sutures.
* Subjects are followed for 12 months to evaluate outcomes and potential complications.

ELIGIBILITY:
Inclusion Criteria:

Subjects are considered appropriate candidates for the study if they fulfill the following criteria:

1. Subject is willing to give consent and comply with evaluation and treatment schedule;
2. 21 to 60 years of age (inclusive);
3. BMI > 35 kg/m2 and < 50 kg/m2 (BMI 35-40 kg/m2 allowable with one or more significant medical conditions related to obesity, including co-morbid conditions of hyperlipidemia, mild obstructive sleep apnea (per Investigators discretion), hypertension, or osteoarthritis of the hip or knee per investigational site's criteria for which the subject is being treated, and which are generally expected to be improved, reversed, or resolved by weight loss);
4. Candidate for surgical weight loss intervention (i.e., meets ASMBS24 and NIH criteria);
5. Absence of significant psychopathology that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations, per site standard of care (SOC); and
6. Agree to refrain from any type of elective procedures that would affect body weight such as abdominal lipoplasty or liposuction, mammoplasty, or removal of excess skin for the duration of the trial.

Exclusion Criteria:

Subjects will be excluded from the study for any of the following:

1. Women of childbearing potential who are pregnant or lactating at the time of screening or at the time of surgery;
2. Documented history of drug and/or alcohol abuse within two (2) years of the Screening Visit;
3. Previous mal-absorptive or restrictive procedures performed for the treatment of obesity;
4. Scheduled concurrent surgical procedure;
5. Participation in any other investigational device or drug study (non survey based trial) within 12 weeks of enrollment;
6. Any condition which precludes compliance with the study, including:

   1. Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease or ulcerative colitis that have been active within the past 10 years;
   2. Congenital or acquired anomalies of the GI tract, including atresias or stenosis;
   3. Severe cardiopulmonary disease or other serious organic disease that makes the subject a high-risk surgical candidate;
   4. Uncontrolled hypertension;
   5. Portal hypertension;
   6. Treatment with insulin (more than 50 units a day);
   7. Chronic or acute upper gastrointestinal bleeding conditions (e.g., gastric or esophageal varices);
   8. Cirrhosis;
   9. Congenital or acquired intestinal telangiectasia;
   10. Esophageal or gastric disorders including moderate severe preoperative reflux, dysmotility, or Barrett's esophagus;
   11. Presence of hiatal hernia;
   12. Prior surgery of the foregut including hiatal hernia repair or prior gastric surgery;
   13. Pancreatitis;
   14. Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
   15. Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study;
7. History or presence of pre-existing autoimmune connective tissue disease;
8. Use of prescription or over the counter weight reduction medications or supplements within thirty days of the Screening Visit or the duration of study participation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Schauer, M.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period started April 17, 2008. Enrollment continued until December 31, 2008. The followup period continued until January 29, 2010. Enrollment was conducted in the bariatric and research offices of The Cleveland Clinic Foundation, Cleveland, Ohio.
Period: Overall Study
Arm/Group | Anterior Curve | Greater Curve
Started | 9 | 6
Completed | 5 (3 subjects lost to follow up; 1 subject did not complete due to noncompliance of scheduled visits.) | 6
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Noncompliance with scheduled visits. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Curve | Greater Curve | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (10.37) | 36.8 (8.42) | 41.7 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Successful Gastric Plication Using Reduction Gastroplasty
Description: The number of participants who completed the study and had post-opeartive gastrocopies showing intact plications.
Time Frame: Immediately post-operative
Measure: Number; unit: participants
Arm/Group | Anterior Curve | Greater Curve
Number analyzed (Participants) | 9 | 6
participants | 9 | 6

2. Secondary Outcome: Durability of Gastric Plications Following Reduction Gastroplasty
Description: The number of participants who completed month 12 gastroscopies showing intact plications.
Time Frame: 12 month
Population: Includes only participants who completed month 12 gastroscopy.
Measure: Number; unit: participants
Arm/Group | Anterior Curve | Greater Curve
Number analyzed (Participants) | 5 | 6
participants | 4 | 5

3. Secondary Outcome: Weight Loss Following Reduction Gastroplasty
Description: Percentage of excess weight loss calculated at 12 months post-surgery. Percentage of excess weight loss is calculated is the difference in baseline and post-surgery weight divided by the difference in baseline weight and ideal body weight multiplied by 100.
Time Frame: 12 months
Population: Includes only participants who completed month 12 visit.
Measure: Mean (Standard Deviation); unit: Percentage of weight loss
Arm/Group | Anterior Curve | Greater Curve
Number analyzed (Participants) | 5 | 6
Percentage of weight loss | 23.30 (24.88) | 53.43 (22.67)

ADVERSE EVENTS:
Time Frame: 13 months
Description: AEs were collected from the screening visit until the study completion visit at 1 year post surgery.
Arm/Group | Anterior Curve | Greater Curve
Serious Adverse Events (participants affected / at risk) | 0/9 | 2/6
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Curve (N=9) | Greater Curve (N=6)
Acute Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ecessive Post Operative Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Curve (N=9) | Greater Curve (N=6)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 6 (10)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
blood glucose increased (Investigations) | 1 (1) | 0 (0)
blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
chest discomfort (General disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1)
dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
early satiety (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1)
fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
hypertension (Vascular disorders) | 3 (3) | 2 (2)
hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 7 (7) | 6 (7)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
oedema peripheral (General disorders) | 0 (0) | 1 (1)
oral candidiasis (Infections and infestations) | 0 (0) | 1 (2)
pain (General disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
prokeratosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 1 (1)
skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
vision blurred (Eye disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No